CLINICAL TRIAL: NCT04101526
Title: Developing and Testing a Spanish-Language Intervention to Reduce Cancer-Related Sleep Disturbance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-20086
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-Intervention Qualitative Interviews (No Intervention): Qualitative interviews will be conducted with breast cancer survivors, survivors' caregivers, cancer support group leaders and clinicians regarding sleep disturbance in breast cancer survivors and preferences for an intervention for sleep disturbance.
- Videoconference Spanish-language Cognitive-Behavioral Therapy for Insomnia (CBT-I) (Experimental): Behavioral: New Spanish-language Cognitive-Behavioral Therapy for Insomnia (CBT-I) delivered via videoconference
  Interventions: Behavioral: Spanish-language Cognitive-Behavioral Therapy for Insomnia (CBT-I) delivered via videoconference
- Waitlist control group (No Intervention): No intervention until 6 weeks after the baseline assessment, at which point participants complete a follow-up assessment and then are offered the new CBT-I intervention.

INTERVENTIONS:
Behavioral: Spanish-language Cognitive-Behavioral Therapy for Insomnia (CBT-I) delivered via videoconference — Six sessions of Spanish-language Cognitive-Behavioral Therapy for Insomnia (CBT-I) delivered via videoconference. Sessions address topics such as sleep education, sleep hygiene, sleep restriction, stimulus control, relapse prevention, and cognitive restructuring.
  Arms: Videoconference Spanish-language Cognitive-Behavioral Therapy for Insomnia (CBT-I)

SUMMARY:
The purpose of this study is to learn about how to provide treatment to cancer survivors who have difficulty sleeping.

ELIGIBILITY:
Inclusion Criteria:

* Located in the Southern Puerto Rico area
* Able to speak and read Spanish
* Have no documented or observable disabilities that would interfere with study participation
* Has completed primary treatment for breast cancer (e.g., surgery, chemotherapy, radiation)
* Has clinically significant sleep disturbance (i.e., >/= 8 on the Insomnia Severity Index)
* Is at low risk of other sleep disorders that are not amenable to treatment with cognitive-behavioral therapy
* Has access to the Internet and a digital device (e.g., smartphone) capable of using videoconference software

Exclusion Criteria:

* Not able to read and speak Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Gonzalez, PhD, Principal Investigator — H. Lee Moffitt Cancer and Research Institute
Locations (2):
- H Lee Moffitt Cancer and Research Institute, Tampa, Florida, United States
- Ponce Health Services University, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811
- [Derived] Oswald LB, Morales-Cruz J, Eisel SL, Del Rio J, Hoogland AI, Ortiz-Rosado V, Soto-Lopez G, Rodriguez-Rivera E, Savard J, Castro E, Jim HSL, Gonzalez BD. Pilot randomized controlled trial of eHealth cognitive-behavioral therapy for insomnia among Spanish-speaking breast cancer survivors. J Behav Med. 2022 Jun;45(3):503-508. doi: 10.1007/s10865-022-00313-6. Epub 2022 Apr 19. PMID 35438442

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Videoconference Spanish-language Cognitive-Behavioral Therapy for Insomnia (CBT-I) | Waitlist Control Group
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Did not complete all sleep diary entries | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Videoconference Spanish-language Cognitive-Behavioral Therapy for Insomnia (CBT-I) | Waitlist Control Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 24
  >=65 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 15 | 30
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 4 | 6
  More than one race | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate - Acceptability of New Intervention for Cancer-Related Sleep Disturbances
Description: The study will be deemed acceptable if ≥ 50% of eligible cancer survivors who are approached agree to participate. Recruitment rate will be measured by percentage of patients enrolled.
Time Frame: Baseline
Population: 33 eligible candidates were approached for participation in the trial
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Cancer Survivors Who Were Approached Agreed to Participate: Recruitment rates are calculated for all potential study candidates.
Arm/Group | Eligible Cancer Survivors Who Were Approached Agreed to Participate
Number analyzed (Participants) | 33
Participants | 30

2. Primary Outcome: Self Report Outcome - Acceptability of New Intervention for Cancer-Related Sleep Disturbances
Description: The study will be deemed acceptable if > 50% of intervention group participants report that, on average, they agree with positive statements about the intervention (i.e., report an average score of >3 on a scale of 0 to 4).
Time Frame: Approximately 6 weeks after first intervention session
Population: Data was not collected from the participants in the "Wait list Control Group"
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Videoconference Spanish-language Cognitive-Behavioral Therapy for Insomnia (CBT-I)
Number analyzed (Participants) | 15
score on a scale | 3.56 (0.28)

3. Primary Outcome: Number of Participants Attending Educational Component - Feasibility of New Intervention for Cancer-Related Sleep Disturbances
Description: The study will be deemed feasible if ≥ 75% of the intervention group participants attend at least half of the educational components of the intervention. This will be operationalized as having attended at least half of the sessions.
Time Frame: approximately 6 weeks after first intervention session
Population: Data was not collected from the participants in the "Wait list Control Group"
Measure: Count of Participants; unit: Participants
Arm/Group | Videoconference Spanish-language Cognitive-Behavioral Therapy for Insomnia (CBT-I)
Number analyzed (Participants) | 15
Participants | 15

4. Secondary Outcome: Efficacy of New Intervention Using PSQI Scoring
Description: Pittsburgh Sleep Quality Index (PSQI) Scoring:
  Duration of Sleep, Sleep Disturbance, Sleep Latency, Days of Disfunction due to Sleepiness, Sleep Efficiency, Overall Sleep Quality, and Meds Needed to Sleep Response Scale 0 (better) 3 (worse). Total Minimum Score 0 (Better), Total Maximum Score 21 (Worse)
  ≤ 5 = Good Sleep Quality >5 = Poor Sleep Quality
Time Frame: Baseline and approximately 6 weeks after first intervention session
Population: 1 participant in wait list control group did not complete all sleep dairy entries.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Videoconference Spanish-language Cognitive-Behavioral Therapy for Insomnia (CBT-I) | Waitlist Control Group
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 11.60 (3.74) | 11.57 (3.25)
  6 week follow up after intervention: number analyzed (Participants) | 15 | 14
  6 week follow up after intervention | 7.40 (3.25) | 11.77 (3.72)

5. Secondary Outcome: Efficacy of New Intervention Using ISI Scoring
Description: Insomnia Severity Index (ISI) Scoring:
  Sleep Quality, Symptom Severity, Sleep Patterns, Daily Functioning, Insomnia Noticeable to Others, Level of Distress Caused by Insomnia Response Scale 0 (better) 4 (worse) Total Minimum Score 0 (Better) Total Maximum Score 28 (Worse)
  0-7: No Clinically Significant Insomnia 8-14: Subthreshold Insomnia 15-21: Clinical Insomnia 22-28: Severe Clinical Insomnia
Time Frame: Baseline and approximately 6 weeks after first intervention session
Population: 1 participant in wait list control group did not complete all sleep dairy entries.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Videoconference Spanish-language Cognitive-Behavioral Therapy for Insomnia (CBT-I) | Waitlist Control Group
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 18.87 (4.49) | 17.20 (4.49)
  6 week follow up after intervention: number analyzed (Participants) | 15 | 14
  6 week follow up after intervention | 7.80 (3.75) | 13.33 (6.69)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first day of being on study until participant was off study, an average of 6 weeks.
Description: No Adverse Events were reported
Arm/Group | Videoconference Spanish-language Cognitive-Behavioral Therapy for Insomnia (CBT-I) | Waitlist Control Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/26/NCT04101526/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/26/NCT04101526/ICF_000.pdf